CLINICAL TRIAL: NCT01164592
Title: SERVE-HF: Substudy on the Mechanistic Plausibility of the Clinical Benefits of Adaptive Servo-ventilation
Brief Title: Substudy on the Mechanistic Plausibility of the Clinical Benefits of Adaptive Servo-ventilation
Acronym: MS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01a
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Heart Failure; Sleep Disorder; Cheyne Stokes Respiration
Keywords: Heart failure (HF); Sleep disordered breathing (SDB); Cheyne Stokes Respiration (CSR); Adaptive Servoventilation (ASV)
MeSH Terms: conditions — Heart Failure; Sleep Wake Disorders; Cheyne-Stokes Respiration; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapy with adaptive servo ventilation (Active Comparator): optimal medical therapy + adaptive servoventilation
  Interventions: Device: adaptive servoventilation (ASV)
- Optimal medical therapy according to guidelines (No Intervention): optimal medical therapy

INTERVENTIONS:
Device: adaptive servoventilation (ASV) — Patients randomised to therapygroup should use the adaptive servoventilation (ASV) device each night at least 3 hours
  Other Names: Adaptive Servo-Ventilation with AutoSet CS
  Arms: Therapy with adaptive servo ventilation

SUMMARY:
The purpose of this study is to assess changes in left ventricular performance using echocardiography as well as ventricular remodelling, changes in sleep and changes in mood, anxiety and cognitive functions occurring as a result of treatment of predominant central sleep apnoea by adaptive servoventilation (ASV) in chronic heart failure in addition to optimal medical therapy in chronic heart failure. This will be a substudy of the SERVE-HF study.

DETAILED DESCRIPTION:
This substudy is performed within the SERVE-HF Study, a randomised, multi-centre,international trial with parallel group design, with patients randomised to either control (optimal medical management) or active treatment (optimal medical treatment plus use of adaptive servoventilation) in a 1:1 ratio. The randomization will be the same as in the parent study. For this purpose, the randomization of the parent study will be stratified as to whether a patient is included in the substudy or not. 300 patients will be recruited for the substudy overall.

For the purpose of this substudy, patients will be followed up for a period of 12 months.

The following extra tests will be performed at the baseline visit, the 3 months follow up and the 12 months follow up:

* Echocardiogram (for both groups)
* cMRI (for both groups)
* PSG (at the baseline visit only for patients in the treatment group and at 3 months follow up and the 12 months follow up for all patients)
* 4 questionnaires (for both groups)
* Additional blood testing (for both groups)

ELIGIBILITY:
The inclusion and exclusion criteria are mainly those applicable for the parent study; SERVE-HF. The inclusion and exclusion criteria are listed here.

INCLUSION CRITERIA FOR SERVE-HF STUDY:

* Over 22 years of age
* Severe Chronic Heart Failure (CHF) with NYHA class III-IV or NYHA class II with at least one hospitalisation for HF within the last 24 months
* Left ventricular ejection fraction (LVEF) less than or equal to 45% by means of echocardiography, radionucleotide angiography, left ventriculography or cardiac MRI documented less than 12 weeks before randomisation
* Diagnosis of sleep disordered breathing (SDB) with an apnoea-hypopnoea-index (AHI) of >15/hr with at least 50% central events and a central AHI of at least 10/hr
* Clinically stable with no change in medication and no unplanned hospitalisation for heart failure in preceding month
* Optimised medical treatment according to the applicable guidelines
* Able to provide informed consent

ADDITIONAL INCLUSION CRITERIA FOR THE SUBSTUDY

• Predominant central sleep apnoea (apnoea hypopnoea index > 15/hour with ≥ 50% central events and a central AHI ≥10/hour, derived from full polysomnography (based on total sleep time), documented less than 4 weeks before randomization. Flow measurements have to be performed with nasal cannula

EXCLUSION CRITERIA FOR THE SERVE-HF STUDY:

* Significant chronic obstructive pulmonary disease (COPD) with Forced Expiratory Volume within one second (FEV1)<50% predicted
* Oxygen saturation at rest during the day 90% at the time of inclusion
* Current use of Positive Airway Pressure (PAP) therapy
* Life expectancy < 1 year for diseases unrelated to chronic heart failure
* Cardiac surgery, Percutaneous coronary intervention (PCI), Myocardial Infarction (MI) or unstable angina within 6 months prior to randomisation
* Implantation of ICD (implanted cardiodefibrillator) or CRT (cardiac resynchronisation therapy) scheduled or within 6 months prior to randomisation
* Transient ischemic attack (TIA) or Stroke within 3 months prior to randomisation
* Primary hemodynamically significant uncorrected valvular heart disease, obstructive or regurgitant, or any valvular disease expected to lead to surgery during the trial
* Acute myocarditis/pericarditis within 6 months prior to randomisation
* Untreated or therapy refractory Restless legs Syndrome (RLS)
* Pregnancy

ADDITIONAL EXCLUSION CRITERIA FOR THE SUBSTUDY

* Amyloidosis, hypertrophic obstructive cardiomyopathy or arteriovenous fistulas
* Dosage changes of diuretics more than doubled within the last 4 weeks prior to randomisation

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2012-08; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) from baseline to 12 months of therapy as measured by echocardiography (Echo). | Baseline (Randomization), 6- and 12 month-Follow-up-visit

SECONDARY OUTCOMES:
Changes in left and right ventricular function | Baseline (Randomization), 6-and 12-month-Follow-up visit
Changes in LV systolic and diastolic indexed volumes | Baseline (Randomization), 6- and 12-month-Follow-up-visit
Changes in right ventricular (RV) systolic and diastolic indexed volumes | Baseline (Randomization), 6- and 12-month-Follow-up-visit
Changes in LV and RV mass | Baseline (Randomization), 6- and 12-month-Follow-up-visit
Changes in LV sphericity index and LV end-systolic global wall stress | Baseline (Randomization), 6- and 12-month-Follow-up-visit
Changes in sleep duration and sleep stages as well as arousals | Baseline (Randomization), 6- and 12-month-Follow-up-visit
Changes in sleep-disordered breathing | Baseline (Randomization), 6- and 12-month-Follow-up-visit
Changes in quality of life assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline (Randomization), 6- and 12-month-Follow-up-visit
Changes in mental status assessed by Mini-Mental State Examination (MMSE) | Baseline (Randomization), 6- and 12-month-Follow-up-visit
Changes in Patient Health Questionnaire-9 (PHQ-9) score and Patient Anxiety Questionnaire GAD-7 | Baseline (Randomization), 6- and 12-month-Follow-up-visit

CONTACTS AND LOCATIONS:
Overall Officials: Martin Cowie, Prof, Principal Investigator — Royal Brompton Hospital, London; Holger Woehrle, MD, Study Director — ResMed
Locations (94):
- Australia (6):
  - Westmead Hospital, Westmead, New South Wales
  - Rivercity Private Hospital, Auchenflower, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Melbourne Sleep Disorders Centre, East Melbourne, Victoria
  - St. Vincents and Mercy Private Hospital, Melbourne, Victoria
  - Hollywood Private Hospital (CVS), Nedlands, Western Australia
- St. Anne's University Hospital, Brno, Czechia
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Unesta Research Centre, Tampere
  - Tampere University Hospital, Pirkanmaa sairaanhoitopiiri, Tampere
- France (3):
  - Clinique Mutualiste des Eaux Claires, Grenoble
  - CHU Grenoble, Hopital Michallon, Grenoble
  - CHU de Poitiers, Poitiers
- Germany (77):
  - Universitätsklinikum Aachen, Aachen
  - DRK Krankenhaus, Alzey
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Charité Campus Mitte CCM, Berlin
  - Charité Campus Mitte, Berlin
  - POLIKUM Friedenau, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Jüdisches Krankenhaus Berlin, Berlin
  - Praxis für Lunge Herz und Schlaf, Bielefeld
  - Kardiologische Praxis Marschner, Bonn
  - Helios Klinikum Borna, Borna
  - Kardiologie Brühl, Brühl
  - Gemeinschaftspraxis Kardiologie Dr. Becker, Castrop-Rauxel
  - Kardiologische Praxis Dr. Isbruch, Castrop-Rauxel
  - Malteser Krankenhaus St. Hildegardis, Cologne
  - Klinikum der Universität zu Köln- Herzzentrum, Cologne
  - Klinikum der Universität zu Köln-Schlaflabor, Cologne
  - Praxis Dr. Anselm Bäumer, Cologne
  - Gemeinschaftspraxis Dres. Gysan/Heinzler/May, Cologne
  - Praxis Dr. Hecker, Dortmund
  - Kardiologische Praxis Dr. Wetzel, Dortmund
  - Praxis Dr. Lodde, Dortmund
  - Facharztzentrum Dresden-Neustadt GbR, Dresden
  - Gemeinschaftpraxis Dres. Schmidt/Gronke, Dresden
  - Praxis Dr. Hohensee, Dresden
  - Herzzentrum Universität Dresden, Dresden
  - Khs Florence-Nightingale, Düsseldorf
  - Kardiologie Oberkassel, Düsseldorf
  - Gemeinschaftspraxis PD Dr. Lankisch, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Kardiologie Praxis Dr. Bonnekamp, Essen
  - Praxis Dr. Tekiyeh, Essen
  - Ruhrlandklinik Essen, Essen
  - Kath. Kliniken Essen/ Philippusstift, Essen
  - Gemeinschaftspraxis Dres. Guckenbiehl, Flonheim
  - CardioVaskuläres Centrum Frankfurt, Frankfurt
  - Praxis Dr. Diedrichs, Frechen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Kardiologische Praxis Gütersloh, Gütersloh
  - Gemeinschaftspraxis Dres Leischik/Littwitz, Hagen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Lungenklinik Hemer, Hemer
  - B&B GmbH, Herne
  - Cardio-Praxis Herne Dr. Furche, Herne
  - Gemeinschaftspraxis Dr. Bruch, Herne
  - Kardiologische Praxis Dr. Schlichting, Herne
  - Augusta-Kranken-Anstalt gGmbH Thoraxzentrum Ruhrgebiet, Herne
  - St. Elisabeth-Hospital Herten gGmbH, Herten
  - Lungenfachklinik Immenhausen, Immenhausen
  - Cardiopraxis Ingelheim, Ingelheim
  - Gemeinschaftspraxis Dres. Dobler/Turin, Karlstadt am Main
  - Universität Leipzig -Herzzentrum, Leipzig
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck-Kardiologie, Lübeck
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck-Schlaflabor, Lübeck
  - Praxis für Kardiologie Dr. med. Menz, Menden
  - Krankenhaus Bethanien, Moers
  - Kardiologische Praxis Dr. Schön, Mühldorf
  - Evangelisches Krankenhaus Mülheim, Mülheim
  - Lungenärzte am Rotkreuzplatz, München
  - Klinikum Augustinum München, München
  - Universitätsklinikum Münster, Münster
  - Städtisches Khs Lukas, Neuss
  - Kardiologische Praxis Nienburg, Nienburg
  - Praxis Dr. Fröhlich, Ratingen
  - Universitätsklinikum Regensburg, Regensburg
  - Khs St. Adolf Stift, Reinbek
  - Praxis Dr. Hein, Reinbek
  - Katharinen Hospital Unna, Unna
  - Praxis Dr. Gerritsen, Waldkraiburg
  - Kardiologisch angiologische Gemeinschaftspraxis, Wiesbaden
  - Kardiologische Gemeinschaftspraxis Dr. K. Vorbeck, Wiesbaden
  - Missionsärztliche Klinik Würzburg, Würzburg
  - Comprehensive Heart Failure Center, Universitätsklinikum Würzburg, Würzburg
- University Medical Center Groningen, Groningen, Netherlands
- Switzerland (2):
  - Cardiocentro Ticino, Lugano
  - Ospedale Regionale di Lugano, Lugano
- Brompton Hospital, London, London, United Kingdom